CLINICAL TRIAL: NCT05973708
Title: Comparative Effects of Clamshells and Frog Pump Exercises on Gluteus Medius Strengthening and Lower Extremity Function in Runners With Iliotibial Band Syndrome
Brief Title: Comparative Effects of Clamshells and Frog Pump Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0411
Record Dates: First submitted 2023-06-27; First posted 2023-08-03 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Iliotibial Band Syndrome
Keywords: gluteus medius; pain; iliotibial band syndrome; strength
MeSH Terms: conditions — Iliotibial Band Syndrome; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Clamshell Exercise (Active Comparator): Group B will be given frog pumps exercises in their regular training program.
  These exercises are given as:
  * In (0-2) week ,2 sets 10 repetitions
  * In (2-4)week, 3 sets of 10 repetitions
  * In (4-6)week, 3 sets of 15 repetitions
  Interventions: Other: Clamshell Exercise
- Group B: Frog Pump Exercise (Active Comparator): Group B will be given frog pumps exercises in their regular training program.
  These exercises are given as:
  * In (0-2) week ,2 sets 10 repetitions
  * In (2-4)week, 3 sets of 10 repetitions
  * In (4-6)week, 3 sets of 15 repetitions
  Interventions: Other: Frog pump exercise

INTERVENTIONS:
Other: Clamshell Exercise — Clamshell Exercise: The clamshell exercise keeps the hips moving, it strengthens both the gluteus medius AND gluteus maximus. The gluteus medius is the main abductor (movement away from the midline of the body) and external rotator of the hip.
  Arms: Group A: Clamshell Exercise
Other: Frog pump exercise — Frog pump exercise: The frog hip thrust mainly targets the gluteal muscles responsible for thigh extension and abduction. The exercise also works the hamstrings on the back of the thighs which helps in hip extension.
  Arms: Group B: Frog Pump Exercise

SUMMARY:
Iliotibial band syndrome is where a tendon called iliotibial band gets irritated or swollen from rubbing against hip or knee when it gets too tensed. Iliotibial band (ITB) syndrome (ITBS) is the most common cause of lateral knee pain among athletes who are involved in sports that require continuous running or repetitive knee flexion and extension. The incidence ranges from 1.6% to 12% in runners. The aim of the study is to compare the effects of clamshells and frog pump exercises on gluteus medius strengthening and lower extremity function in runners with iliotibial band syndrome.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial and will be conducted in Pakistan Sports Board Lahore. Non-probability convenient sampling will be used to collect the data. Sample size of 32 subjects with age group between 18-30 years (males) will be taken. Data will be collected from the runners with tight ITB, by using tools LEFS, HOS-SS, and Hand held dynamometer. An informed consent will be taken. A total of 26 subjects will be selected by following inclusion and exclusion criteria and will equally divided in to two groups by random number generator table. Both the Groups will continue the conventional training with Group A will receive clamshell Exercise, and Group B will receive frog pump exercise in their respective training programs. Outcome measures will be measured at baseline and after 2 weeks. Data analysis will be done by SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* • Age (18-30yrs)

  * Gender (Males)
  * Positive Ober's test
  * Positive Noble's compression test
  * Suffering pain from past 3 months
  * Running approximately 5km/week

Exclusion Criteria:

* • Osteoporosis

  * Previous knee trauma/surgery
  * Patellofemoral joint pain
  * Popliteus tendinitis
  * Lateral meniscal injure

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Manual Muscle Testing (MMT) | upto 6th weeks
  For measuring the strength of Hip muscles, Manual Muscle Testing (MMT) is used.
  Manual Muscle Testing (MMT) is a standardised set of assessments that measure muscle strength and function against specific criteria and is commonly used in clinical practice by physiotherapists.
  Grading Scale Range: 0 to 5 0 None No visible or palpable contraction
  1. Trace Visible or palpable contraction with no motion
  2. Poor Full ROM gravity eliminated
  3. Fair Full ROM against gravity
  4. Good Full ROM against gravity, moderate resistance
  5. Normal Full ROM against gravity, maximum resistance
Hip Outcome Score (HOS) | upto 6th weeks
  The hip outcome score (HOS) is a questionnaire used to measure the function of the Hip.
  The HOS is a patient-completed measure that consists of an "Activities of Daily Living" subscale (17 scored items) and a "Sports" subscale (9 scored items) in which the response options are presented as 5-point Likert scales (Scores 0-4).
Lower Extremity Functional Scale (LEFS) | upto 6th weeks
  The lower extremity functional scale (LEFS) measures the function and disability of the lower extremity.
  LEFS is a well-known and validated instrument for the measurement of lower extremity function. The LEFS was developed in a group of patients with various musculoskeletal disorders.
  The LEFS rating scale categories are: (1) "extreme difficulty or unable to perform," (2) "quite a bit of difficulty," (3) "moderate difficulty," (4) "a little bit of difficulty," and (5) "no difficulty." LEFS score = SUM (points for all 20 activities) Interpretation: Minimum score: 0 Maximum score: 80 The lower the score the greater the disability.

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, Mphil, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Pakistan Sports Board, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friede MC, Innerhofer G, Fink C, Alegre LM, Csapo R. Conservative treatment of iliotibial band syndrome in runners: Are we targeting the right goals? Phys Ther Sport. 2022 Mar;54:44-52. doi: 10.1016/j.ptsp.2021.12.006. Epub 2021 Dec 27. PMID 35007886
- [Background] Baker RL, Souza RB, Fredericson M. Iliotibial band syndrome: soft tissue and biomechanical factors in evaluation and treatment. PM R. 2011 Jun;3(6):550-61. doi: 10.1016/j.pmrj.2011.01.002. PMID 21665168
- [Background] Khaund R, Flynn SH. Iliotibial band syndrome: a common source of knee pain. Am Fam Physician. 2005 Apr 15;71(8):1545-50. PMID 15864895
- [Background] Fredericson M, Guillet M, Debenedictis L. Innovative solutions for iliotibial band syndrome. Phys Sportsmed. 2000 Feb;28(2):53-68. doi: 10.3810/psm.2000.02.693. PMID 20086621
- [Background] McKay J, Maffulli N, Aicale R, Taunton J. Iliotibial band syndrome rehabilitation in female runners: a pilot randomized study. J Orthop Surg Res. 2020 May 24;15(1):188. doi: 10.1186/s13018-020-01713-7. PMID 32448384
- [Background] Fredericson M, Wolf C. Iliotibial band syndrome in runners: innovations in treatment. Sports Med. 2005;35(5):451-9. doi: 10.2165/00007256-200535050-00006. PMID 15896092